CLINICAL TRIAL: NCT06161623
Title: The Effect of Laughter Yoga Applied to Intensive Care Nurses on Perceived Stress, Work Motivation, and Mental Well-Being
Brief Title: The Effect of Laughter Yoga on Perceived Stress, Work Motivation, and Mental Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCBU-K-CEVIK-002
Record Dates: First submitted 2023-11-04; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Mental Health; Complementary Therapies
Keywords: Laughter yoga; Perceived stress; Work motivation; Mental well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Yoga Application (Experimental): The intervention group took eight sessions of laughter yoga, that is, two sessions per week for 4 weeks. The participants in the intervention group were asked to fill in the data collection tools before the laughter yoga sessions, and after the 4th and 8th yoga sessions
  Interventions: Behavioral: Laughter Yoga Application
- Control group (No Intervention): The participants in the control group also filled in the data collection tools without undergoing any intervention.

INTERVENTIONS:
Behavioral: Laughter Yoga Application — The intervention group took eight sessions of laughter yoga, that is, two sessions per week for 4 weeks. The participants in the intervention group were asked to fill in the data collection tools before the laughter yoga sessions, and after the 4th and 8th yoga sessions.
  Arms: Laughter Yoga Application

SUMMARY:
The aim of this randomized controlled experimental study is to examine the effect of laughter yoga applied to intensive care nurses on perceived stress, work motivation, and mental well-being.

DETAILED DESCRIPTION:
The study was conducted with nurses working at Manisa Celal Bayar University Hospital's Surgical Intensive Care and Anesthesia Intensive Care units between December 2022 and March 2023. The Nurse Introduction Form, Nurse Work Motivation Scale, Perceived Stress Scale, and Warwick-Edinburgh Mental Well-being Scale were used to collect data.

ELIGIBILITY:
Inclusion Criteria: Between 18-65 age

* Those who have worked as intensive care nurses for at least 6 months
* Those who agree to participate in the research

Exclusion Criteria:

* Those with chronic cough
* Those who have previously received laughter yoga training and practiced
* Those who had surgery within the last 3 months
* Those with diagnosed mental illness and those using medication (antidepressants, antipsychotics,anxiolytic, etc…)
* Those who have neurological diseases such as epilepsy and multiple sclerosis
* Those who have recently experienced a loss (within at least 6 months)
* Those with neurological disorders
* Those who have urinary incontinence problems
* Those who did not agree to participate in the research

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Work Motivation | 2 weeks
  Work Motivation Scale was used. The highest score the scale can get in total is 75, while the lowest score is 25.
  High scale scores mean that nurses have high work motivation.
Perceived Stress | 2 weeks
  Perceived Stress Scale was used. A high total score on the scale indicates that the individual perceives high stress.
  High scores on the subscales are generally interpreted as negative.
Mental Well-being | 2 weeks
  Warwick-Edinburgh Mental Well-being Scale was used. It can score between a minimum of 14 and a maximum of 70 points.
  High scores indicate that the individual is in a good psychological state.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Yılmaz, Principal Investigator — Celal Bayar University
Locations (1):
- Kivan Çevik Kaya, Manisa, MANİSAYunusemre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will be given if it's necessary and if it is not problem for ethical office.